CLINICAL TRIAL: NCT03505190
Title: A Randomized, Sponsor-Open, Investigator-Blind, Subject-Blind, Placebo-Controlled, Single Ascending Dose, to Investigate the Safety, Tolerability and Pharmacokinetics of RO7062931 Following Subcutaneously Administration in Healthy Chinese Volunteers
Brief Title: A Study to Evaluate the Safety, Tolerability and Pharmacokinetics of RO7062931 in Healthy Chinese Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: YP39432
Record Dates: First submitted 2018-04-13; First posted 2018-04-23 (Actual); Results first posted 2020-08-03 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Healthy Participants
MeSH Terms: interventions — RO7062931

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- RO7062931 0.3mg/kg (Experimental): Participants will receive subcutaneously (SC) 0.3 milligram per kilogram (mg/kg) of RO7062931.
  Interventions: Drug: RO7062931; Drug: Placebo
- RO7062931 1.0mg/kg (Experimental): Participants will receive subcutaneously (SC) 1.0 milligram per kilogram (mg/kg) of RO7062931.
  Interventions: Drug: RO7062931; Drug: Placebo
- RO7062931 2.0mg/kg (Experimental): Participants will receive subcutaneously (SC) 2.0 milligram per kilogram (mg/kg) of RO7062931.
  Interventions: Drug: RO7062931; Drug: Placebo
- RO7062931 4.0mg/kg (Experimental): Participants will receive subcutaneously (SC) 4.0 milligram per kilogram (mg/kg) of RO7062931.
  Interventions: Drug: RO7062931; Drug: Placebo
- Placebo (Placebo Comparator): Participants will receive matching placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RO7062931 — RO7062931 will be administered SC in single ascending doses with starting of 0.3 mg/kg and subsequent doses of 1.0 mg/kg, 2.0 mg/kg and 3.0 mg/kg, respectively. Additional (optional) dose of 4.0 mg/kg may be administered based on safety, tolerability and PK data.
  Arms: RO7062931 0.3mg/kg; RO7062931 1.0mg/kg; RO7062931 2.0mg/kg; RO7062931 4.0mg/kg
Drug: Placebo — Matching placebo will be administered subcutaneously (SC).

SUMMARY:
This randomized study will evaluate the safety, tolerability and pharmacokinetics of single ascending subcutaneously administered doses of RO7062931 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Chinese healthy male and female (of non-childbearing potential) volunteers.
* A Body Mass Index (BMI) between 19 to 27 kilogram per square meter (kg/m2) inclusive and a body weight of at least 45 kg.
* Women should be of non-childbearing potential. These include those who have undergone surgical sterilization (removal of ovaries and/or uterus) or are post-menopausal.
* Men must agree to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures during treatment and up to 105 days after the last dose of RO7062931, and agree to refrain from donating sperm during this same period.
* Non-smoker (nor tobacco containing products) for at least 90 days prior to dosing on Day 1 and agree to remain as non-smoker during the study.

Exclusion Criteria:

* History of drug or alcohol abuse or dependence in previous 6 months.
* Positive urine drug and alcohol screen or positive cotinine test at Screening or Day -1.
* Positive result on hepatitis B (HBV), hepatitis C (HCV), or human immunodeficiency virus (HIV)-1 and -2 at Screening.
* Confirmed blood pressure or resting pulse rate outside of accepted ranges.
* Participation in an investigational drug or device study within 90 days prior to screening.
* Donation of blood over 500 milliliters (mL) within three months prior to screening.
* Any major illness within the one month, or any febrile illness within two weeks preceding the screening visit.
* Alcohol consumption of more than 2 standard drinks per day on average.
* Screening or baseline ECG evidence of atrial fibrillation, atrial flutter, complete right or left bundle branch block, Wolff-Parkinson-White syndrome, or cardiac pacemaker.
* Any out of range findings in liver function tests, INR and renal function tests or any clinically significant abnormalities (as judged by the Investigator) in the physical examination and in the remaining laboratory test results (including hepatic and renal panels, complete blood count, chemistry panel and urinalysis) at Screening or on Day-1.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2019-07-05 (Actual); Study Completion 2019-07-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong
  - Prince of Wales Hospital, Shatin, New Territories

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Planned: Up to 50 healthy volunteers (HVs) across 5 cohorts of 10 HVs (8 active, 2 placebo) per dose-level.
  Actual: A total of 41 HVs were enrolled across 4 dose cohorts.
Period: Overall Study
Arm/Group | RO7062931 0.3mg/kg | RO7062931 1.0mg/kg | RO7062931 2.0mg/kg | RO7062931 4.0mg/kg | Placebo
Started | 9 | 8 | 8 | 8 | 8
Completed | 9 | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RO7062931 0.3mg/kg | RO7062931 1.0mg/kg | RO7062931 2.0mg/kg | RO7062931 4.0mg/kg | Placebo | Total
Number analyzed (Participants) | 9 | 8 | 8 | 8 | 8 | 41
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.8 (6.4) | 29.3 (11.5) | 29.8 (11.0) | 29.6 (9.2) | 34.5 (15.) | 30.2 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 9 | 8 | 8 | 8 | 8 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 8 | 8 | 8 | 8 | 41
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian/ Chinese | 9 | 8 | 8 | 8 | 8 | 41

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events and AEs of Special Interest
Description: Adverse events of special interest for this study include the following:
  * Cases of an elevated ALT or AST in combination with either an elevated bilirubin or clinical jaundice
  * Suspected transmission of an infectious agent by the study drug
  * Severe injection site reactions
  * Renal adverse events
Time Frame: Up to 16 weeks
Population: The Safety Population was defined as all Healthy Volunteers who have received at least one dose of the study medication, whether prematurely withdrawn from the study or not.
Measure: Number; unit: Percentage of Participants
Arm/Group | RO7062931 0.3mg/kg | RO7062931 1.0mg/kg | RO7062931 2.0mg/kg | RO7062931 4.0mg/kg | Placebo
Number analyzed (Participants) | 9 | 8 | 8 | 8 | 8
Percentage of Participants
  Adverse Events | 66.7 | 62.5 | 62.5 | 75.0 | 87.5
  Adverse Events of Special interest (AESI) | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Percentage of Participants With Marked Laboratory Abnormalities Based on Hematology, Blood Chemistry, Coagulation and Urinalysis Test Results
Description: Marked reference range has been predefined for each laboratory parameter. The marked reference range is broader than the standard reference range. Values falling outside the marked reference range that also represent a defined change from baseline will be considered marked laboratory abnormalities (i.e., potentially clinically relevant). If a baseline value is not available for a study subject, the midpoint of the standard reference range will be used as the study participant baseline value for the purposes of determining marked laboratory abnormalities.
Time Frame: Baseline, Day 2, 8, 15, 29, 85
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | RO7062931 0.3mg/kg | RO7062931 1.0mg/kg | RO7062931 2.0mg/kg | RO7062931 4.0mg/kg | Placebo
Number analyzed (Participants) | 9 | 8 | 8 | 8 | 8
Percentage of Participants
  SGOT/AST High | 11.1 | 0 | 0 | 0 | 0
  Neutrophils, Total, Abs, Low | 0 | 0 | 12.5 | 0 | 0
  Triglycerides High | 0 | 0 | 12.5 | 0 | 12.5

3. Primary Outcome: Percentage of Participants With Electrocardiogram (ECG) Abnormalities
Description: Table entries provide the percentage of Participants with a during treatment assessment abnormality in the direction specified regardless of this abnormality at baseline. Abnormalities reported in Participants with missing baseline values are included. Baseline is the Participant's last observation prior to initiation of study drug.
Time Frame: Baseline; pre-dose, 1 hour (h), 4, 8, 12h post-dose Day 1, 24h post-dose Day 2, 8, 15, 29, 85
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | RO7062931 0.3mg/kg | RO7062931 1.0mg/kg | RO7062931 2.0mg/kg | RO7062931 4.0mg/kg | Placebo
Number analyzed (Participants) | 9 | 8 | 8 | 8 | 8
Percentage of Participants
  Heart Rate Low | 0 | 0 | 0 | 0 | 0
  Heart Rate High | 0 | 0 | 0 | 0 | 0
  PR Duration Low | 11.1 | 0 | 0 | 0 | 12.5
  PR Duration High | 0 | 25.0 | 0 | 0 | 25.0
  QRS Duration Low | 0 | 0 | 0 | 0 | 0
  QRS Duration High | 0 | 0 | 0 | 0 | 0
  QT Duration Low | 0 | 0 | 0 | 0 | 0
  QT Duration High | 0 | 0 | 0 | 0 | 0
  QTcF - Fridericia's Correction Formula Low | 0 | 12.5 | 0 | 0 | 0
  QTcF - Fridericia's Correction Formula High | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Maximum Plasma Concentration (Cmax) for RO7062931
Description: Observed Maximum Plasma Concentration were obtained after the participants received the RO7062931
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 18h post-dose Day 1, 24, 30, 36h post-dose Day 2, Day 3, 4, 5, 6, 8
Population: The PK analysis population included all healthy volunteers randomized and adherent to the protocol. Participants were excluded if they significantly violated the inclusion/exclusion criteria, deviated significantly from the protocol or if data were unavailable or incomplete. Data presented is only for participants included in the actual analysis
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | RO7062931 0.3mg/kg | RO7062931 1.0mg/kg | RO7062931 2.0mg/kg | RO7062931 4.0mg/kg | Placebo
Number analyzed (Participants) | 9 | 8 | 8 | 8 | 0
nmol/L | 17.71 (39.5) | 57.09 (28.8) | 113.52 (40.3) | 299.39 (36.5) |

5. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) for RO7062931
Description: Time to reach the observed Maximum Plasma Concentration were obtained after the participants received the RO7062931.
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 18h post-dose Day 1, 24, 30, 36h post-dose Day 2, Day 3, 4, 5, 6, 8
Population: as for outcome 4
Measure: Median (Full Range); unit: h
Arm/Group | RO7062931 0.3mg/kg | RO7062931 1.0mg/kg | RO7062931 2.0mg/kg | RO7062931 4.0mg/kg | Placebo
Number analyzed (Participants) | 9 | 8 | 8 | 8 | 0
h | 1.50 [1.0 to 3.0] | 2.38 [1.0 to 3.9] | 2.87 [1.9 to 3.9] | 2.85 [1.4 to 4.0] |

6. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinity (AUC0-inf) for RO7062931
Description: Area Under the Plasma Concentration-time Curve Extrapolated to infinity was calculated based on Non-Compartment Analysis.
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 18h post-dose Day 1, 24, 30, 36h post-dose Day 2, Day 3, 4, 5, 6, 8
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*nmol/L
Arm/Group | RO7062931 0.3mg/kg | RO7062931 1.0mg/kg | RO7062931 2.0mg/kg | RO7062931 4.0mg/kg | Placebo
Number analyzed (Participants) | 9 | 8 | 8 | 8 | 0
h*nmol/L | 95.26 (9.0) | 349.75 (14.8) | 791.99 (19.9) | 2180.74 (8.3) |

7. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero Until the Last Quantifiable Time-Point (AUC0-last) for RO7062931
Description: Area Under the Plasma Concentration-time Curve up to the last measurable concentration was calculated based on Non-Compartment Analysis
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 18h post-dose Day 1, 24, 30, 36h post-dose Day 2, Day 3, 4, 5, 6, 8
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*nmol/L
Arm/Group | RO7062931 0.3mg/kg | RO7062931 1.0mg/kg | RO7062931 2.0mg/kg | RO7062931 4.0mg/kg | Placebo
Number analyzed (Participants) | 9 | 8 | 8 | 8 | 0
h*nmol/L | 95.16 (9.0) | 348.33 (14.8) | 786.33 (20.8) | 2114.90 (10.9) |

8. Secondary Outcome: Terminal Elimination Half-Life (t1/2) for RO7062931
Description: Terminal Half-life was calculated based on Non-Compartment Analysis.
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 18h post-dose Day 1, 24, 30, 36h post-dose Day 2, Day 3, 4, 5, 6, 8
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | RO7062931 0.3mg/kg | RO7062931 1.0mg/kg | RO7062931 2.0mg/kg | RO7062931 4.0mg/kg | Placebo
Number analyzed (Participants) | 9 | 8 | 8 | 8 | 0
h | 3.87 (44.6) | 66.59 (38.6) | 81.83 (24.0) | 88.78 (18.4) |

9. Secondary Outcome: Apparent Clearance (CL/F) for RO7062931
Description: Apparent oral clearance was calculated from Dose/AUCinf.
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 18h post-dose Day 1, 24, 30, 36h post-dose Day 2, Day 3, 4, 5, 6, 8
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | RO7062931 0.3mg/kg | RO7062931 1.0mg/kg | RO7062931 2.0mg/kg | RO7062931 4.0mg/kg | Placebo
Number analyzed (Participants) | 9 | 8 | 8 | 8 | 0
L/h | 29.24 (11.4) | 27.23 (18.8) | 25.24 (18.5) | 17.46 (8.4) |

10. Secondary Outcome: Apparent Volume of Distribution (Vz/F) for RO7062931
Description: Apparent volume of distribution was calculated from Dose/AUCinf
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 18h post-dose Day 1, 24, 30, 36h post-dose Day 2, Day 3, 4, 5, 6, 8
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | RO7062931 0.3mg/kg | RO7062931 1.0mg/kg | RO7062931 2.0mg/kg | RO7062931 4.0mg/kg | Placebo
Number analyzed (Participants) | 9 | 8 | 8 | 8 | 0
L | 163.27 (45.7) | 2616.31 (35.8) | 2980.22 (40.0) | 2235.97 (15.3) |

11. Secondary Outcome: Cumulative Amount of RO7062931 Excreted in Urine (Ae)
Description: Ae: cumulative amount of drug excreted in urine over a 24 hour period or over defined time periods linked to the pools of urine collected.
Time Frame: (0-4), (4-8), (8-12), (12-24)h post-dose Day 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: nmol
Arm/Group | RO7062931 0.3mg/kg | RO7062931 1.0mg/kg | RO7062931 2.0mg/kg | RO7062931 4.0mg/kg | Placebo
Number analyzed (Participants) | 9 | 8 | 8 | 8 | 0
nmol
  Ae 0-8h | 35.35 (6.64) | 133.79 (29.09) | 326.90 (106.77) | 1433.92 (595.77) |
  Ae 0-24h | 41.88 (6.69) | 147.88 (40.78) | 545.61 (139.56) | 1977.71 (513.27) |

12. Secondary Outcome: Fraction of Cumulative Amount of RO7062931 Excreted in the Urine Over Total Dose (Fe)
Description: The fraction of cumulative amount in urine were calculated based on Ae/Dose
Time Frame: 0-24h h post-dose Day 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | RO7062931 0.3mg/kg | RO7062931 1.0mg/kg | RO7062931 2.0mg/kg | RO7062931 4.0mg/kg | Placebo
Number analyzed (Participants) | 9 | 8 | 8 | 8 | 0
Percentage | 1.50 (0.20) | 1.63 (0.30) | 2.79 (0.72) | 5.26 (1.65) |

13. Primary Outcome: Percentage of Participants With T-wave Abnormalities
Description: as for outcome 3
Time Frame: Baseline; pre-dose, 1 hour (h), 4, 8, 12h post-dose Day 1, 24h post-dose Day 2, 8, 15, 29, 85
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | RO7062931 0.3mg/kg | RO7062931 1.0mg/kg | RO7062931 2.0mg/kg | RO7062931 4.0mg/kg | Placebo
Number analyzed (Participants) | 9 | 8 | 8 | 8 | 8
Percentage of Participants
  Baseline Normal | 0 | 0 | 0 | 0 | 0
  Day 1 / 1H | 0 | 0 | 0 | 0 | 0
  Day 1 / 4H | 0 | 0 | 0 | 0 | 0
  Day 1 / 8H | 0 | 0 | 0 | 0 | 0
  Day 1 / 12H | 0 | 0 | 0 | 0 | 0
  Day 2 / 24H | 0 | 0 | 0 | 0 | 0
  Day 8 / 168H | 0 | 0 | 0 | 0 | 0
  Follow-up Visit Day 15 | 0 | 0 | 0 | 0 | 0
  Follow-up Visit Day 29 | 0 | 0 | 0 | 0 | 0
  Follow-up Visit Day 85 | 0 | 0 | 0 | 0 | 0

14. Primary Outcome: Percentage of Participants With U-wave Abnormalities
Description: as for outcome 3
Time Frame: Baseline; pre-dose, 1 hour (h), 4, 8, 12h post-dose Day 1, 24h post-dose Day 2, 8, 15, 29, 85
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | RO7062931 0.3mg/kg | RO7062931 1.0mg/kg | RO7062931 2.0mg/kg | RO7062931 4.0mg/kg | Placebo
Number analyzed (Participants) | 9 | 8 | 8 | 8 | 8
Percentage of Participants
  Baseline Normal | 22.2 | 0 | 0 | 25.0 | 0
  Day 1 / 1H | 11.1 | 0 | 0 | 25.0 | 0
  Day 1 / 4H | 22.2 | 0 | 0 | 0 | 12.5
  Day 1 / 8H | 22.2 | 0 | 0 | 0 | 12.5
  Day 1 / 12H | 22.2 | 0 | 0 | 0 | 12.5
  Day 2 / 24H | 11.1 | 0 | 0 | 0 | 12.5
  Day 8 / 168H | 12.5 | 0 | 0 | 0 | 12.5
  Follow-up Visit Day 15 | 11.1 | 0 | 0 | 12.5 | 0
  Follow-up Visit Day 29 | 0 | 0 | 0 | 0 | 0
  Follow-up Visit Day 85 | 11.1 | 0 | 0 | 12.5 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 14 months
Description: Number of events includes all occurrences. The Safety Population includes all participants who received study drug or placebo.
Arm/Group | RO7062931 0.3mg/kg | RO7062931 1.0mg/kg | RO7062931 2.0mg/kg | RO7062931 4.0mg/kg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/8 | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 6/9 | 5/8 | 5/8 | 6/8 | 7/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RO7062931 0.3mg/kg (N=9) | RO7062931 1.0mg/kg (N=8) | RO7062931 2.0mg/kg (N=8) | RO7062931 4.0mg/kg (N=8) | Placebo (N=8)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Noninfective gingivitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tongue cyst (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site bruise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Injection site reaction (General disorders) | 0 (0) | 2 (2) | 1 (1) | 4 (5) | 1 (1)
Vessel puncture site bruise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vessel puncture site erythema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site pruritus (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 3 (3)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Injection related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-29): https://cdn.clinicaltrials.gov/large-docs/90/NCT03505190/Prot_SAP_000.pdf